CLINICAL TRIAL: NCT03245476
Title: Physiotherapy in Adhesive Capsulitis Pathology: Effect of an Education Based Approach on Arthroscopic Evaluation Results, Joint Range of Motion, Psychosocial Factors, Shoulder Pain and Arm Function
Brief Title: Education-based Physical Therapy Approach for Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Annick Timmermans, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.08/REVA17.01
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Adhesive Capsulitis
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: corticoid injection + physiotherapy with a focus on manual therapy and home-exercises versus corticosteroid injection + physiotherapy with focus on education and supported home exercises
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy and home-exercises (Active Comparator): corticoid injection + physiotherapy with a focus on manual therapy and home-exercises
  Interventions: Other: Physical therapy focus on manual therapy and home-exercises
- education and supported home exercises (Active Comparator): corticosteroid injection + physiotherapy with focus on education and supported home exercises
  Interventions: Other: Physical therapy focus on education and supported home exercises

INTERVENTIONS:
Other: Physical therapy focus on manual therapy and home-exercises — corticoid injection + physiotherapy with a focus on manual therapy and home-exercises
  Arms: manual therapy and home-exercises
Other: Physical therapy focus on education and supported home exercises — corticosteroid injection + physiotherapy with focus on education and supported home exercises
  Arms: education and supported home exercises

SUMMARY:
This study aims, by means of a randomized control trial, to investigate which treatment method (corticoid injection + physiotherapy with a focus on manual therapy and home-exercises versus corticosteroid injection + physiotherapy with focus on education and supported home exercises) gives better results on clinically relevant outcomes (range of glenohumeral motion, psychological factors, pain, shoulder function, quality of life) and on parameters derived from arthroscopic glenohumeral investigation by means of MRI.

Furthermore, associations between (1) the results on the MRI investigation, (2) the range of glenohumeral motion, (3) shoulder function and pain, and (4) psychological factors will be assessed at different time-points (before and at 6-12-18 and 52 weeks after the first injection).

ELIGIBILITY:
Inclusion Criteria:

* 50 % loss of passive GH external rotation motion, together with motion losses greater than 25% in at least two other GH movements, as compared to the unaffected side
* the pain accompanying the motion losses has to be present for at least one month. During that month, the pain and mobility deficits have to be stable or get worse

Exclusion Criteria:

* bilateral frozen shoulder
* systemic and/or neurologic disease or a self-reported pathologic condition of the cervical/thoracic region, elbow or wrist/hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-09-04 (Estimated); Primary Completion 2019-09-04 (Estimated); Study Completion 2019-09-04 (Estimated)

PRIMARY OUTCOMES:
Scapulothoracic, glenohumeral and elbow joint range of motion | baseline
  before the first injection with corticosteroids By means of inertial motion sensors, range of motion in the scapulothoracic, glenohumeral and elbow joint will be assessed during functional task performance
Scapulothoracic, glenohumeral and elbow joint range of motion | week 6
  after the first injection with corticosteroids. By means of inertial motion sensors, range of motion in the scapulothoracic, glenohumeral and elbow joint will be assessed during functional task performance
Scapulothoracic, glenohumeral and elbow joint range of motion | week 12
  after the first injection with corticosteroids. By means of inertial motion sensors, range of motion in the scapulothoracic, glenohumeral and elbow joint will be assessed during functional task performance
Scapulothoracic, glenohumeral and elbow joint range of motion | week 18
  after the first injection with corticosteroids. By means of inertial motion sensors, range of motion in the scapulothoracic, glenohumeral and elbow joint will be assessed during functional task performance
Scapulothoracic, glenohumeral and elbow joint range of motion | week 52
  after the first injection with corticosteroids. By means of inertial motion sensors, range of motion in the scapulothoracic, glenohumeral and elbow joint will be assessed during functional task performance
parameters on arthrographic investigation by means of MRI | baseline
  the thickness of the coracohumeral ligament, the capacity of the inferior glenohumeral joint recessus are investigated.
parameters on arthrographic investigation by means of MRI | week 18
  the thickness of the coracohumeral ligament, the capacity of the inferior glenohumeral joint recessus are investigated.
Disability of the shoulder, elbow and hand questionnaire | baseline
  assessment of upper limb function
Disability of the shoulder, elbow and hand questionnaire | week 6
  assessment of upper limb function
Disability of the shoulder, elbow and hand questionnaire | week 12
  assessment of upper limb function
Disability of the shoulder, elbow and hand questionnaire | week 18
  assessment of upper limb function
Disability of the shoulder, elbow and hand questionnaire | week 52
  assessment of upper limb function
Brief pain inventory | baseline
  assessment of current, worst and night pain on a 11 point likert scale
Brief pain inventory | week 6
  assessment of current, worst and night pain on a 11 point likert scale
Brief pain inventory | week 12
  assessment of current, worst and night pain on a 11 point likert scale
Brief pain inventory | week 18
  assessment of current, worst and night pain on a 11 point likert scale
Brief pain inventory | week 52
  assessment of current, worst and night pain on a 11 point likert scale

SECONDARY OUTCOMES:
EQ-5D-5L questionnaire | baseline
  Quality of life assessment
EQ-5D-5L questionnaire | week 6
  Quality of life assessment
EQ-5D-5L questionnaire | week 12
  Quality of life assessment
EQ-5D-5L questionnaire | week 18
  Quality of life assessment
EQ-5D-5L questionnaire | week 52
  Quality of life assessment
Self-efficacy questionnaire | baseline
  this questionnaire assesses the self-efficacy of a person
Self-efficacy questionnaire | week 6
  this questionnaire assesses the self-efficacy of a person
Self-efficacy questionnaire | week 12
  this questionnaire assesses the self-efficacy of a person
Self-efficacy questionnaire | week 18
  this questionnaire assesses the self-efficacy of a person
Self-efficacy questionnaire | week 52
  this questionnaire assesses the self-efficacy of a person
Tampa scale of kinesiophobia | baseline
  this scale investigates fear of movement
Tampa scale of kinesiophobia | week 6
  this scale investigates fear of movement
Tampa scale of kinesiophobia | week 12
  this scale investigates fear of movement
Tampa scale of kinesiophobia | week 18
  this scale investigates fear of movement
Tampa scale of kinesiophobia | week 52
  this scale investigates fear of movement
Hospital anxiety and depression scale | baseline
  this scale investigates anxiety and depression
Hospital anxiety and depression scale | week 6
  this scale investigates anxiety and depression
Hospital anxiety and depression scale | week 12
  this scale investigates anxiety and depression
Hospital anxiety and depression scale | week 18
  this scale investigates anxiety and depression
Hospital anxiety and depression scale | week 52
  this scale investigates anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Liesbet De Baets, dr., Study Chair — Hasselt University; Annick Timmermans, prof. dr., Principal Investigator — Hasselt University; Carl Dierickx, prof. dr., Study Chair — Jessa ziekenhuis, Universiteit Hasselt
Locations (1):
- Jessa Ziekenhuis, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: Undecided